CLINICAL TRIAL: NCT04538612
Title: DiCART TM Device for Capillary Refill Time Measurement : a Validation Study.
Brief Title: DiCART TM Device for Capillary Refill Time Measurement
Acronym: DICART-VS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL18_0217; 2019-A00094-53 (Other: IDRCB)
Record Dates: First submitted 2020-08-28; First posted 2020-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Perfusion
Keywords: capillary refill time; vascular occlusion test; device; impaired perfusion; healthy volunteers.

STUDY DESIGN:
Masking Description: the investigators evaluate capillary refill time without knowing the status of vascular occlusion test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- measure capillary refill time (Experimental)
  Interventions: Device: measure capillary refill time

INTERVENTIONS:
Device: measure capillary refill time — Each time, capillary refill time will be evaluated three times consecutively by clinical method applying a firm pressure with the finger during 15s, then brutally releasing it, and estimating time of skin recoloration with a chronometer and by DiCART TM device
  Three vascular occlusion tests will be successively performed with a cuff during less than 10 minutes:
  * Arterial vascular occlusion test (50mmHg above systolic arterial pressure of the healthy volunteers),
  * Veinous vascular occlusion test (30mmHg),
  * Control test without vascular occlusion test. Capillary refill time measurements will be repeated just before, during and just after vascular occlusion tests.
  Randomization determine the order of the vascular occlusion tests. Investigators performing capillary refill time evaluation will be blinded from it. Vascular occlusion tests will be alternatively performed by one and the other limb. The whole protocol will be performed at the upper and then at the lower limb.

SUMMARY:
To estimate peripheral perfusion in shock state, international guidelines recommend the use of capillary refill time, and practitioners currently evaluates it at bedside. However its measurement is not standardized, what should explain the large observer variability reported in different studies. Hence, a device providing a standardized evaluation seems to be helpful.

The aim of the study is to evaluate diagnostic performance of such a device recently developped (DiCART TM), in healthy volunteers experiencing vascular occlusion tests to induce impaired perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age > 18 years old
* Informed consent to participate

Exclusion Criteria:

* Vascular disease
* Diabetes mellitus
* Dermatosis
* Cutaneous lesion on a measurement site
* Anemia
* Pregnancy
* Cardiovascular chronic treatment
* Non affiliation to a social security regime
* Involvement in other interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Capillary refill time on the thenar eminence evaluated with DiCART TM device. | 180 minutes
  Diagnostic performance of DiCART TM device to detect a capillary refill time variation on the thenar eminence induced by a vascular occlusion test on the arm.
  DiCART TM measurement is fully automatized, and may be separated in three consecutive step :
  * An automatized cutaneous compression
  * A video acquisition of cutaneous recoloration
  * Data interpretation The investigators will compute Receptor Operative Characteristics curves with area under the curve, and will determine best threshold and grey zone to evaluate diagnostic performance of DiCART TM device to detect impaired perfusion.

SECONDARY OUTCOMES:
Capillary refill time evaluated on the knee with DiCART TM device | 180 minutes
  Diagnostic performance of DiCART TM device to detect a capillary refill time variation on the knee induced by a vascular occlusion test on the leg
  DiCART TM measurement is fully automatized, and may be separated in three consecutive step :
  * An automatized cutaneous compression
  * A video acquisition of cutaneous recoloration
  * Data interpretation The investigators will compute Receptor Operative Characteristics curves with area under the curve, and will determine best threshold and grey zone to evaluate diagnostic performance of DiCART TM device to detect impaired perfusion.
Intra -observer variability of capillary refill time measurement with DiCART TM device by performing repetitive measurements by two different investigators. | 180 minutes
  Two different investigators will realize 5 measurements of capillary refill time with DiCART TM device and standard clinical method in physiological conditions in two different sites (knee and thenar eminence). We will compute least significant change and standard deviation/mean ratio to evaluate observer variability.
Intra -observer variability of capillary refill time measurement with clinical method by performing repetitive measurements by two different investigators. | 180 minutes
  Two different investigators will realize 5 measurements of capillary refill time with DiCART TM device and standard clinical method in physiological conditions in two different sites (knee and thenar eminence). We will compute least significant change and standard deviation/mean ratio to evaluate observer variability.
Inter-observer variability of capillary refill time measurement with DiCART TM device by performing repetitive measurements by two different investigators. | 180 minutes
  Two different investigators will realize 5 measurements of capillary refill time with DiCART TM device and standard clinical method in physiological conditions in two different sites (knee and thenar eminence). We will compute least significant change and standard deviation/mean ratio to evaluate observer variability.
Inter-observer variability of capillary refill time measurement with clinical method by performing repetitive measurements by two different investigators. | 180 minutes
  Two different investigators will realize 5 measurements of capillary refill time with DiCART TM device and standard clinical method in physiological conditions in two different sites (knee and thenar eminence). We will compute least significant change and standard deviation/mean ratio to evaluate observer variability.
Capillary refill time variation induced by vascular occlusion test on the knee with DiCART TM device | 180 minutes
  Standard clinical measurement is realized by applying a firm pressure with the finger during 15s and by brutally releasing it. Then, skin recoloration is evaluated visually with a chronometer.
Capillary refill time variation induced by vascular occlusion test on the knee with standard clinical method | 180 minutes
  Standard clinical measurement is realized by applying a firm pressure with the finger during 15s and by brutally releasing it. Then, skin recoloration is evaluated visually with a chronometer.
Capillary refill time variation induced by vascular occlusion test on the thenar eminence with DiCART TM device . | 180 minutes
  Standard clinical measurement is realized by applying a firm pressure with the finger during 15s and by brutally releasing it. Then, skin recoloration is evaluated visually with a chronometer.
Capillary refill time variation induced by vascular occlusion test on the thenar eminence with standard clinical method. | 180 minutes
  Standard clinical measurement is realized by applying a firm pressure with the finger during 15s and by brutally releasing it. Then, skin recoloration is evaluated visually with a chronometer.
Capillary refill time measured by mathematical algorithms | 180 minutes
  After the experimental phase, the investigators will develop mathematical algorithms to optimize video data interpretation.
number of patients with cutaneous lesions | 180 minutes
  To evaluate the safety of DiCART TM device
Pain evaluation assessed by numeric rating scale | 180 minutes
  Pain scale (minimum 1 to maximum 10), 1=No pain,10=Unbearable pain

CONTACTS AND LOCATIONS:
Overall Officials: Matthias JACQUET-LAGREZE, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospital Louis Pradel, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ruste M, Cazenave L, Tardif M, Saint-Jean C, Fellahi JL, Lagreze MJ. Measurement of capillary refill time with a handheld prototype device: a comparative validation study in healthy volunteers. J Clin Monit Comput. 2022 Oct;36(5):1271-1278. doi: 10.1007/s10877-021-00757-2. Epub 2021 Sep 22. PMID 34550528